CLINICAL TRIAL: NCT02906137
Title: Altered Homing of T Lymphocytes to the Gut and Poor Immune Reconstitution of the Intestinal Mucosa in Treated HIV-infected Individuals
Brief Title: Gut-Associated Lymphocyte Trafficking
Acronym: GALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANRS EP61 GALT
Record Dates: First submitted 2016-08-17; First posted 2016-09-19 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-1 infected subjects (Experimental): 40 subjects will be recruited in the Department of Infectious Diseases of Toulouse University Hospital, France:
  * 15 subjects will have an upper endoscopy (gastroscopy) with duodenal sampling
  * 15 subjects will have a lower endoscopy (coloscopy) with colonic and ileal sampling
  * 10 subjects will have both a gastroscopy and a coloscopy
  Interventions: Other: Peripheral blood and intestinal biopsies will be collected
- Uninfected-controls (Other): 40 subjects will be recruited in the Department of Internal Medicine of Toulouse University Hospital, France:
  * 10 subjects will have an upper endoscopy (gastroscopy) with duodenal sampling
  * 10 subjects will have a lower endoscopy (coloscopy) with colonic and ileal sampling
  * 20 subjects will have both a gastroscopy and a coloscopy
  Interventions: Other: Peripheral blood and intestinal biopsies will be collected

INTERVENTIONS:
Other: Peripheral blood and intestinal biopsies will be collected — Blood draw and intestinal biopsies

SUMMARY:
The gut immune barrier is not fully restored in HIV-1-infected subjects despite they were receiving antiretroviral treatment. This leaky gut leads to microbial translocation from the gut lumen into the bloodstream that fuels deleterious systemic inflammation. The chemotaxis axes that allow T lymphocytes to migrate from the blood to the gut mucosa in order to reconstitute the mucosal immune barrier seems altered in treated HIV-1-infected subjects.This study aims at better understanding the mechanisms involved in this lack of mucosal immune restoration.

DETAILED DESCRIPTION:
Pathophysiological study in human subjects, comparative, national, multicentric and prospective. Peripheral blood and intestinal biopsies will be collected.

ELIGIBILITY:
Inclusion Criteria are:

For HIV-1-infected subjects group :

* Age at least 18-year old
* HIV-1 infection
* Receiving continuous cART for ≥ 12 months, started during the chronic phase
* Plasma viral load ≤50 copies/mL for ≥ 6 months (one blip ≤200 copies/mL authorized)
* Blood CD4+ T cells count ≥ 350 cells/mm3
* Indication for upper and/or lower digestive endoscopy
* Patient enrolled in or a beneficiary of a Social Security programme (State Medical Aid or AME is not a Social Security programme)
* Written informed consent.

For uninfected control group :

* Age at least 18-year old
* Indication for upper and/or lower digestive endoscopy
* Patient enrolled in or a beneficiary of a Social Security programme (State Medical Aid or AME is not a Social Security programme)
* Written informed consent

Exclusion Criteria are:

For HIV-1-infected subject group :

* HIV-2 infection
* Inflammatory bowel diseases (Crohn's disease, ulcerative colitis) ; coeliac disease
* Platelets count <50 G/L or abnormal hemostasis tests
* Decompensated cirrhosis
* Past or current lymphoma
* Involvement in an HIV-1 immunotherapeutic vaccine study
* Pregnant or breastfeeding women
* Subjects participating in a study excluding participating in another study
* Vulnerability, such as an age under 18, tutorship, trusteeship, or subjects deprived of liberty by a legal or administrative decision.

For uninfected control group :

* HIV-1 and 2 infection
* Inflammatory bowel diseases (Crohn's disease, ulcerative colitis) ; coeliac disease
* Platelets count <50 G/L or abnormal hemostasis tests
* Decompensated cirrhosis
* Past or current lymphoma
* Pregnant or breastfeeding women
* Subjects participating in a study excluding participating in another study
* Vulnerability, such as an age under 18, tutorship, trusteeship, or subjects deprived of liberty by a legal or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Immune status: Measure of the frequencies of Th1 in peripheral blood and gut mucosa. | Baseline
  The frequencies of Th1 will be measured by flow cytometry.
Immune status: Measure of the frequencies of Th17 in peripheral blood and gut mucosa. | Baseline
  The frequencies of Th17 will be measured by flow cytometry.
Immune status: Measure of the frequencies of Th22 in peripheral blood and gut mucosa. | Baseline
  The frequencies of Th22 will be measured by flow cytometry.

SECONDARY OUTCOMES:
Immune status: Quantification of cytokines in blood and gut mucosa. | Baseline
  The quantification of cytokines will be measured by luminex.
Immune status: Quantification of cytokines in blood and gut mucosa. | Baseline
  The quantification of cytokines will be measured by immuno-histochemistry.
Immune status: Quantification of chemiokines in blood and gut mucosa. | Baseline
  The quantification of chemiokines will be measured by luminex.
Immune status: Quantification of chemiokines in blood and gut mucosa. | Baseline
  The quantification of chemiokines will be measured by immuno-histochemistry.
Microbial translocation : Quantification of soluble CD14 in plasma. | Baseline
  The quantification of CD 14 will be realised by Enzyme-Linked Immunosorbent Assay (ELISA).
Microbial translocation : Quantification of soluble soluble CD163 in plasma. | Baseline
  The quantification of CD163 will be realised by Enzyme-Linked Immunosorbent Assay (ELISA) .
Microbial translocation : Quantification of Lipopolysaccharide Binding Protein (LBP). | Baseline
  The quantification of Lipopolysaccharide Binding Protein will be realised by Enzyme-Linked Immunosorbent Assay (ELISA).
Microbial translocation : Quantification of Intestinal-type Fatty Acid-Binding Protein (I-FABP) in plasma. | Baseline
  The quantification of Intestinal-type Fatty Acid-Binding Protein (I-FABP) will be realised by Enzyme-Linked Immunosorbent Assay (ELISA).
Microbial translocation : Quantification of 16S RNA. | Baseline
  The quantification of 16S RNA will be realised by real-time Polymerase Chaine Reaction (qPCR).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Purpan - Service de Médecine Interne, Toulouse
  - Hôpital Purpan - Service des maladies Infectieuses, Toulouse

IPD SHARING:
Plan to Share IPD: No